CLINICAL TRIAL: NCT07203950
Title: Effectiveness of Global Postural Reeducation on Psychophysical Wellbeing in Housewives With Chronic Non-specific Low Back Pain
Brief Title: Effects of Global Postural Reeducation on Psychophysical Wellbeing in Housewives With Chronic Non-specific LBP.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/F24C08G30004 Roha Farooqi
Record Dates: First submitted 2025-09-25; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Low Back Pain; Stress; Sleep Quality
Keywords: low back pain; stress; sleep quality; global postural reeducation
MeSH Terms: conditions — Low Back Pain; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Global Postural Reeducation (Experimental): Participants assigned to this arm will undergo Global Postural Reeducation (GPR) using standardized coxofemoral positions ( Opening and Closing). In the Opening position, the participant lies supine with the hip placed in gentle flexion, abduction, and external rotation to lengthen the medial/anterior muscle chain; in the Closing position, the hip is positioned in slight extension, adduction, and internal rotation to target the lateral/posterior chain. Each session lasts approximately 10 minutes, divided into 2-3 blocks of 3-5 minutes each, during which participants perform slow diaphragmatic breathing combined with gentle isometric contractions (2-3 seconds) on exhalation followed by relaxation into the posture. Sessions are delivered twice weekly for 6 weeks. Therapist monitoring ensures proper pelvic stabilization, safe range of motion, and avoidance of compensatory movements, while participants are encouraged to maintain comfortable stretch intensity without pain.
  Interventions: Other: global postural reeducation with conventional therapy
- Conventional Therapy (Active Comparator): * Hot pack for 15 minutes.
  * Static stretching of rectus femoris and iliopsoas muscles (1 minute x 5 repetitions per session).
  * Other exercises Pelvic tilt Straight leg raise Bridging Cat-camel exercise Knee-to-chest stretch Prescribed as 3 sets of 10 repetitions each, with rest in between.
  Interventions: Other: conventional therapy

INTERVENTIONS:
Other: global postural reeducation with conventional therapy — Global postural reeducation will include two postural positions aiming to improve alignment, flexibility and postural correction. Each session will be 35 minutes including each posture performed for 10 minutes each and 15 minutes for conventional therapy.
  1. Coxofemoral Opening with Closed Arms Participants will begin in a supine position on a flat surface. The upper limbs will be 90° abducted, with palms facing to the ceiling. The lower limbs will be placed in hip and knee flexion, with soles of the feet together, heels close to the gluteal region, and hips in abduction between 30° and 45°.
  2. Coxofemoral Closure with Closed Arms. In this posture, participants will again lie supine, with the arms abducted to 90° and palms facing upward. The hips and knees will be flexed, with the soles of the feet pressed together and placed against a wall.
     with Controlled and slow diaphragmatic breathing technique
  3. Conventional therapy same as given to other group.
  Arms: Global Postural Reeducation
Other: conventional therapy — conventional therapy given to this group will be
  * Hot pack for 15 minutes.
  * Static stretching of rectus femoris and iliopsoas muscles (1 minute x 5 repetitions per session).
  * Other exercises Pelvic tilt Straight leg raise Bridging Cat-camel exercise Knee-to-chest stretch Prescribed as 3 sets of 10 repetitions each, with rest in between.
  Arms: Conventional Therapy

SUMMARY:
This study aims to explore the multidimensional impact of Global postural reeducation in a population that is not only physically overburdened but also psychologically strained due to the demands of domestic life. Unlike conventional therapies that often focus solely on pain relief, GPR offers a comprehensive intervention model that may simultaneously enhance physical function, reduce psychological stress, and improve sleep quality. By targeting housewives with chronic non-specific LBP, this study seeks to fill a critical gap in the literature and provide evidence for a more inclusive, preventive, and non-pharmacological approach to musculoskeletal and mental health management

DETAILED DESCRIPTION:
Low back Pain (LBP) is a primary cause of disability among people of all ages and a major contributor to the global burden of diseases. Non-specific low back pain is a form of low back pain without any specific identified underlying disease or any anatomical abnormality. Global postural reeducation (GPR) is a physical therapy protocol that focuses on eccentrically stretching the muscular chains which are shortened due to behavioral, psychological and constitutional factors. For this method physical therapists guide the patients a series of gentle active movements and maintain postures aiming to stretch the shortened muscles, realign the joints and also enhance the contraction of antagonist muscles. It is a randomized control trial which will be conducted on 30 patients calculated using G*power software. Patients fulfilling the inclusion criteria will be randomized into 2 groups i.e. GROUP A (global postural reeducation with conventional therapy) & GROUP B (conventional therapy). Patients in Group A will receive global postural reeducation technique with conventional therapy and Group B will receive conventional therapy alone which includes hot pack for 15 minutes, Static stretching for iliopsoas and rectus femoris and other exercises two times a week.

Outcomes will be measured at baseline and at the end of 3rd week, at the end of 6th week.

ELIGIBILITY:
Inclusion Criteria:

Participants' full filling the criteria given below will be recruited in this study. Diagnosis based on clinical guidelines linked to the International Classiﬁcation of Function, Disability and Health of the Orthopedic Section of the American Physiotherapy Association.

1. Housewives (Age 25-40 years)
2. Chronic nonspecific LBP (more than 3 months)
3. Experience mild to moderate stress (measured by perceived stress scale)
4. Sleep disturbances or poor sleep quality (PSQI score>5)

Exclusion Criteria:

Participant falling in this category would be excluded of the study.

1. Pregnancy.
2. Using NSAIDs.
3. Acute, subacute LBP.
4. Females having diagnosed irregular/prolonged menstrual cycles.
5. History of recent Spinal surgery (within the past year).
6. Neurological deficits (foot drop, motor weakness).
7. Diagnosed severe psychiatric issues (e.g. severe depression, bipolar disorder, psychosis).
8. Use of sleep medications, antidepressants, or anxiolytics during the study period.
9. Specific causes of LBP (herniated disc, lumbar stenosis, spinal deformity, fracture, spondolysthesis).
10. Systemic diseases (tumor, Rhematoid arthritis)

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
numeric pain rating scale | Assessed at Baseline, 3 weeks, and 6-week follow-up.
  The NPRS is an 11-point self-report scale ranging from 0 (no pain) to 10 (worst imaginable pain). Participants are asked to rate their average pain intensity in the lower back during daily activities over the past 24 hours.
lumber ROMs using inclinometer | Assessed at Baseline, 3 weeks, and 6-week follow-up.
  Lumbar spine mobility will be assessed in flexion, extension, lateral flexion, and rotation using a digital inclinometer. The inclinometer will be placed at standardized anatomical landmarks (spinous process of T12 and sacrum for flexion/extension; along midline for lateral flexion/rotation).
perceived stress scale | Assessed at Baseline, 3 weeks, and 6-week follow-up.
  The PSS-10 is a 10-item validated questionnaire that measures the degree to which participants perceive situations in their life as stressful over the past month. Items assess feelings of unpredictability, lack of control, and overload.
Pittsburg sleep quality index | Assessed at Baseline, 3 weeks, and 6-week follow-up.
  The PSQI is a 19-item validated questionnaire assessing subjective sleep quality and disturbances over the past month. It generates 7 component scores (sleep duration, disturbance, latency, efficiency, quality, medication use, and daytime dysfunction).

CONTACTS AND LOCATIONS:
Overall Officials: Ramsha Tariq, MSPT(OMPT), Principal Investigator — Riphah International University
Locations (1):
- Dr Zushmaleen Ahmed Chughtai Physiotherapy Clinic, Kot Addu, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Watanabe M, Tomiyama C, Nikaido T, Takeda T, Mandai N. Mental status is significantly associated with low back pain: a survey-based cross-sectional study among Japanese women. BMC Res Notes. 2023 Jan 30;16(1):8. doi: 10.1186/s13104-023-06276-4. PMID 36717870
- [Background] Gonzalez-Medina G, Perez-Cabezas V, Ruiz-Molinero C, Chamorro-Moriana G, Jimenez-Rejano JJ, Galan-Mercant A. Effectiveness of Global Postural Re-Education in Chronic Non-Specific Low Back Pain: Systematic Review and Meta-Analysis. J Clin Med. 2021 Nov 16;10(22):5327. doi: 10.3390/jcm10225327. PMID 34830609
- [Background] Kandil EA, Yamany AAER, Alsaka SSD, Abd El-Azeim AS. Effect of global postural reeducation on chronic low pain patients with lower cross syndrome. Bulletin of Faculty of Physical Therapy. 2024;29(1):8.
- [Background] Rodriguez-Aragon M, Varillas-Delgado D, Gordo-Herrera J, Fernandez-Ezequiel A, Moreno-Heredero B, Valle N. Effects of global postural re-education on stress and sleep quality in health sciences female students: a randomized controlled trial pilot study. Front Psychiatry. 2024 Aug 28;15:1404544. doi: 10.3389/fpsyt.2024.1404544. eCollection 2024. PMID 39262580
- [Background] Rodriguez-Aragon M, Barranco-Rodriguez D, de Mora-Martin M, Sanchez-Jorge S, Varillas-Delgado D, Valle-Benitez N. The effects of global postural re-education on sleep quality and stress in university women lecturers: a randomized controlled trial. Front Psychiatry. 2024 Jan 16;14:1321588. doi: 10.3389/fpsyt.2023.1321588. eCollection 2023. PMID 38298929